CLINICAL TRIAL: NCT00150449
Title: A 1-Year Open-Label Safety Extension Study of Pregabalin in Patients With Anxiety Disorders
Brief Title: Determine Long-Term Safety and Tolerability of Pregabalin in Patients With Anxiety Disorders.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1008-100
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2006-07-14 (Estimated); Status verified 2006-07

CONDITIONS: Anxiety Neuroses
MeSH Terms: conditions — Anxiety Disorders | interventions — Pregabalin

INTERVENTIONS:
Drug: Pregabalin

SUMMARY:
Determine long-term safety and tolerability of pregabalin in patients with anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* Must have completed the double-blind portion of the preceding trial
* Completed any protocol specified withdrawal phase and follow-up visits.

Exclusion Criteria:

* Patient cannot participate if they experienced a serious adverse event or a nonserious, but medically significant adverse event during the preceding efficacy study that was judged to be related to the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511
Dates: Start 2001-01; Study Completion 2006-03

PRIMARY OUTCOMES:
Safety Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (123):
- Austria (3):
  - Pfizer Investigational Site, A-1040 Wien
  - Pfizer Investigational Site, Vienna
  - Pfizer Investigational Site, Wein
- Belgium (9):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, De Pinte
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Kortrijk
  - Pfizer Investigational Site, Lede
  - Pfizer Investigational Site, Liège
  - Pfizer Investigational Site, Sint-Denijs-Westrem
  - Pfizer Investigational Site, Tielt
  - Pfizer Investigational Site, Tournai
- Estonia (2):
  - Pfizer Investigational Site, Tallinn
  - Pfizer Investigational Site, Tartu
- France (8):
  - Pfizer Investigational Site, Reims, Cedex
  - Pfizer Investigational Site, Denguin
  - Pfizer Investigational Site, Élancourt
  - Pfizer Investigational Site, Metz
  - Pfizer Investigational Site, Montesson
  - Pfizer Investigational Site, Montigny-lès-Metz
  - Pfizer Investigational Site, Saint-Étienne-du-Grès
  - Pfizer Investigational Site, Wasquehal
- Germany (10):
  - Pfizer Investigational Site, Bad-Deurrheim
  - Pfizer Investigational Site, Bremerhaven
  - Pfizer Investigational Site, Göttingen
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Köthen
  - Pfizer Investigational Site, Lauf
  - Pfizer Investigational Site, Oldenburg
  - Pfizer Investigational Site, Osnabrück
  - Pfizer Investigational Site, Siegen
  - Pfizer Investigational Site, Spaichingen
- Pfizer Investigational Site, Ness Ziona, Israel
- Italy (4):
  - Pfizer Investigational Site, Bassano Del Grappa (Vicenza)
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Roma
- Pfizer Investigational Site, Riga, Latvia
- Netherlands (10):
  - Pfizer Investigational Site, BV Losser
  - Pfizer Investigational Site, GC Nijmegen
  - Pfizer Investigational Site, Hoogvliet
  - Pfizer Investigational Site, Huizen
  - Pfizer Investigational Site, Losser
  - Pfizer Investigational Site, RC Dordrecht
  - Pfizer Investigational Site, Vlaardinger-Ambacht
  - Pfizer Investigational Site, Zwigndrecht
  - Pfizer Investigational Site, Zwijndreacht
  - Pfizer Investigational Site, Zwijndrecht
- Poland (9):
  - Pfizer Investigational Site, Bialystok
  - Pfizer Investigational Site, Bydgoszcz
  - Pfizer Investigational Site, Katowice
  - Pfizer Investigational Site, Olsztyn
  - Pfizer Investigational Site, Torun
  - Pfizer Investigational Site, Tuszyn
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
  - Pfizer Investigational Site, Zabrze
- South Africa (16):
  - Pfizer Investigational Site, Goodwood, Cape Town
  - Pfizer Investigational Site, Paarl, Cape Town
  - Pfizer Investigational Site, Kempton Park, Johannesburg
  - Pfizer Investigational Site, Rosebank, Johannesburg
  - Pfizer Investigational Site, Hatfield, Pretoria
  - Pfizer Investigational Site, Bellville
  - Pfizer Investigational Site, Bloemfontein
  - Pfizer Investigational Site, East London
  - Pfizer Investigational Site, George
  - Pfizer Investigational Site, Hurlingham, Johannesburg
  - Pfizer Investigational Site, Pinetown Natal
  - Pfizer Investigational Site, Polokwane
  - Pfizer Investigational Site, Pretoria
  - Pfizer Investigational Site, Sandton
  - Pfizer Investigational Site, Somerset West
  - Pfizer Investigational Site, Westville
- Spain (7):
  - Pfizer Investigational Site, Granollers, Barcelona
  - Pfizer Investigational Site, Oviedo, Principality of Asturias
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Pamplona
  - Pfizer Investigational Site, Seville
  - Pfizer Investigational Site, Zaragoza
- Ukraine (3):
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Lviv
  - Pfizer Investigational Site, Odesa
- United Kingdom (39):
  - Pfizer Investigational Site, Maidenhead, Berkshire
  - Pfizer Investigational Site, Slough, Berks
  - Pfizer Investigational Site, Falmouth, Cornwall
  - Pfizer Investigational Site, Fowey, Cornwall
  - Pfizer Investigational Site, Penzance, CORNWALL
  - Pfizer Investigational Site, Saltash, Cornwall
  - Pfizer Investigational Site, St Austell, CORNWALL
  - Pfizer Investigational Site, Downpatrick, County Down
  - Pfizer Investigational Site, Chesterfield, Derbyshire
  - Pfizer Investigational Site, Plymouth, Devon
  - Pfizer Investigational Site, Bexhill-on-Sea, EAST SUSSEX
  - Pfizer Investigational Site, Bexhill-on-Sea, East Sussex
  - Pfizer Investigational Site, Leigh-on-Sea, Essex
  - Pfizer Investigational Site, Leslie, Fife
  - Pfizer Investigational Site, Limekilns, Fife
  - Pfizer Investigational Site, Cathcart, Glasgow
  - Pfizer Investigational Site, Clarckston, Glasgow
  - Pfizer Investigational Site, Rutherglen, Glasgow
  - Pfizer Investigational Site, Bolton, Lancashire
  - Pfizer Investigational Site, Chelsea, London
  - Pfizer Investigational Site, Bangor, Northern Ireland
  - Pfizer Investigational Site, Greenisland, Carrickfergus, Northern Ireland
  - Pfizer Investigational Site, Houston, Renfrewshire
  - Pfizer Investigational Site, Epworth, Doncaster, South Yorkshire
  - Pfizer Investigational Site, Saint John's, Woking, Surrey
  - Pfizer Investigational Site, Trowbridge, WILTSHIRE
  - Pfizer Investigational Site, Inkberrow, Worcestershire
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, Bolton
  - Pfizer Investigational Site, Chesterfield
  - Pfizer Investigational Site, Cookstown
  - Pfizer Investigational Site, Coventry
  - Pfizer Investigational Site, Dundee
  - Pfizer Investigational Site, Earlsdon, Coventry
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Leeds
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Port Glasgow
  - Pfizer Investigational Site, Rugby
- Pfizer Investigational Site

REFERENCES:
- [Derived] Montgomery S, Emir B, Haswell H, Prieto R. Long-term treatment of anxiety disorders with pregabalin: a 1 year open-label study of safety and tolerability. Curr Med Res Opin. 2013 Oct;29(10):1223-30. doi: 10.1185/03007995.2013.820694. Epub 2013 Aug 19. PMID 23808960
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=1008-100&StudyName=Determine+Long%2DTerm+Safety+and+Tolerability+of+Pregabalin+in+Patients+with+Anxiety+Disorders%2E